CLINICAL TRIAL: NCT00596635
Title: Cranberry for UTI Prevention in Residents of Long Term Care Facilities
Acronym: PACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0606001581; DF06-005
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Results first posted 2010-09-23 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Urinary Tract Infection
Keywords: UTI; elderly; prevention; cranberry; E.Coli
MeSH Terms: conditions — Urinary Tract Infections; Escherichia coli Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Group (No Intervention): No cranberry capsules administered
- One cranberry capsule (Active Comparator): 1 650mg cranberry capsule daily
  Interventions: Dietary Supplement: Once Daily Cranberry Capsule
- Two cranberry capsules (Active Comparator): 1 650 mg cranberry capsule twice daily (bid)
  Interventions: Dietary Supplement: Twice Daily Cranberry Capsules

INTERVENTIONS:
Dietary Supplement: Once Daily Cranberry Capsule — 650mg capsule pure cranberry powder
  Other Names: Theralogix: Theracran cranberry supplement, 650mg capsule
  Arms: One cranberry capsule
Dietary Supplement: Twice Daily Cranberry Capsules — One 650mg cranberry capsule administered twice per day
  Other Names: Theralogix: Theracran cranberry supplement, 650mg capsule
  Arms: Two cranberry capsules

SUMMARY:
Urinary tract infections (UTIs) affect over 7 million men and women per year and cost the health care industry over 1 billion dollars annually. The incidence of UTI increases markedly in elderly institutionalized persons and leads to excessive antimicrobial usage, emergency room visits, hospitalization, sepsis, and death. The use of antimicrobials to prevent UTI in elderly nursing home patients is not recommended and is fraught with problems such as adverse reactions, drug interactions, and the development of drug-resistant organisms. There is no accepted method of preventing UTI in residents of nursing homes, a vulnerable and understudied population with significant morbidity from UTI.

The overall goal of this proposal is to conduct a prospective cohort pilot study that evaluates the feasibility of using cranberry to prevent UTI in nursing home residents. Each of the aims is critical for the optimal design of a larger placebo-controlled, definitive trial of cranberry for prevention of UTI in nursing home residents and will provide the essential preliminary data for future larger studies.

DETAILED DESCRIPTION:
Cranberry products represent a novel, non-antimicrobial method for prevention of UTI. There is evidence for a plausible mechanism and efficacy for UTI prevention in healthy premenopausal women. Limited clinical studies of cranberry products in elderly men and women have demonstrated reductions in bacteriuria but have not been of adequate size or quality to support the use of cranberry in this population or result in changes in patient care. Thus, a properly designed, definitive study demonstrating efficacy of cranberry in preventing UTI in this population is needed. However, before a large-scale, placebo-controlled trial can be justified, the complexities inherent to studying older nursing home residents need to be addressed. These include issues related to collecting uncontaminated urine samples, understanding the microbiology of UTI in this population, and devising an acceptable intervention regimen. The overall goal of this proposal is to conduct a prospective cohort pilot study that evaluates the feasibility of using cranberry to prevent UTI in nursing home residents. Each of the aims listed below is critical for the optimal design of a larger placebo-controlled, definitive trial of cranberry for prevention of UTI in nursing home residents and will provide the essential preliminary data for a future RO1 level grant application.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 60 years old and a resident of the nursing home or assisted living facility for greater than 30 days duration

Exclusion Criteria:

* Having a known major anatomic abnormality of the urinary tract
* Presence of acute UTI symptom
* Intolerance or allergy to cranberry products
* Current use of cranberry for prevention of UTI
* Use of warfarin
* History of kidney stones
* Presence of a chronic indwelling bladder catheter
* Dialysis dependence
* Chronic suppressive antibiotics
* Immunocompromised state due to hematological malignancies, HIV infection, chronic high dose (>10mg daily) prednisone or equivalent steroid use.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Juthani-Mehta, MD, Principal Investigator — Yale University School of Medicine, Assistant Professor
Locations (1):
- Yale University School of Medicine, Internal Medicine, Section of Infectious Diseases, New Haven, Connecticut, United States

REFERENCES:
- [Result] Juthani-Mehta M, Perley L, Chen S, Dziura J, Gupta K. Feasibility of cranberry capsule administration and clean-catch urine collection in long-term care residents. J Am Geriatr Soc. 2010 Oct;58(10):2028-30. doi: 10.1111/j.1532-5415.2010.03080.x. No abstract available. PMID 20929476
- [Derived] Williams G, Stothart CI, Hahn D, Stephens JH, Craig JC, Hodson EM. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2023 Nov 10;11(11):CD001321. doi: 10.1002/14651858.CD001321.pub7. PMID 37947276
- [Derived] Williams G, Hahn D, Stephens JH, Craig JC, Hodson EM. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2023 Apr 17;4(4):CD001321. doi: 10.1002/14651858.CD001321.pub6. PMID 37068952

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four dementia units participated in this study. Exclusion criteria included: 1)indwelling catheter, 2)residence <4 weeks, 3)prednisone therapy, 4)active UTI symptoms, 5)terminal, 6)end stage renal disease, 7)<60 years old, 8)chronic suppressive antibiotic therapy, 9)history of kidney stones, 10)unable to provide baseline urine, 11)warfarin therapy.
Pre-assignment Details: If a participant could not provide a baseline urine specimen or met an exclusion criterion prior to group assignment but after consent, he or she was not enrolled.
Groups:
- No Cranberry Capsules: Control Group No Cranberry Capsule
- 2 Cranberry Capsules: 1 650 mg cranberry capsule twice daily (bid)
Period: Overall Study
Arm/Group | No Cranberry Capsules | One Cranberry Capsule | 2 Cranberry Capsules
Started | 17 | 20 | 19
Completed | 10 | 7 | 11
Not Completed | 7 | 13 | 8
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Treatment for symptomatic UTI | 4 | 6 | 3
Not completed — Hip fracture | 2 | 3 | 3
Not completed — Could not provide urine specimen | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Cranberry Capsules | One Cranberry Capsule | 2 Cranberry Capsules | Total
Number analyzed (Participants) | 17 | 20 | 19 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 0 | 1
  >=65 years | 16 | 20 | 19 | 55
Age Continuous [Mean (Standard Deviation); unit: years] | 85.76 (11.76) | 88.30 (6.16) | 86.68 (5.16) | 86.82 (7.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 16 | 46
  Male | 4 | 3 | 3 | 10
Region of Enrollment [Number; unit: participants]
  United States | 17 | 20 | 19 | 56

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With E.Coli Isolated From Urine Culture
Description: Urine cultures were obtained at baseline and monthly for six months. Any participant that had E.coli isolated at least once is listed as meeting the outcome.
Time Frame: 6 months
Measure: Number; unit: Participants
Arm/Group | No Cranberry Capsules | One Cranberry Capsule | 2 Cranberry Capsules
Number analyzed (Participants) | 17 | 20 | 19
Participants | 8 | 8 | 12

2. Secondary Outcome: Number of Participants With >100,000 Colony Forming Units Per Milliliter of Any Organism Isolated From Urine Culture
Description: Urine cultures were obtained at baseline and monthly for 6 months. If a urine culture had >100,000 colony forming units per milliliter of any organism on any of the urine cultures obtained, the participant is noted as meeting the outcome.
Time Frame: 6 months
Measure: Number; unit: Participants
Arm/Group | No Cranberry Capsules | One Cranberry Capsule | 2 Cranberry Capsules
Number analyzed (Participants) | 17 | 20 | 19
Participants | 12 | 13 | 14

3. Primary Outcome: Number of Urine Cultures Collected Out of the Total Number Expected to be Collected.
Description: Urine cultures were collected at baseline and monthly for six months. The total number of urine cultures collected out of the total number that were expected to be collected are shown.
Time Frame: 6 months
Measure: Number; unit: Urine cultures
Arm/Group | No Cranberry Capsules | One Cranberry Capsule | 2 Cranberry Capsules
Number analyzed (Participants) | 17 | 20 | 19
Urine cultures
  Number of urine cultures expected | 81 | 74 | 85
  Number of urine cultures collected | 73 | 63 | 71

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | No Cranberry Capsules | One Cranberry Capsule | 2 Cranberry Capsules
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 3/17 | 5/20 | 3/19
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Cranberry Capsules (N=17) | One Cranberry Capsule (N=20) | 2 Cranberry Capsules (N=19)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The inability to follow all participants for the full six months reflects the vulnerability of the population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes